CLINICAL TRIAL: NCT05170789
Title: A Phase II, Single-Arm, Study of Elotuzumab, Selinexor, and Dexamethasone in Patients With Relapsed Refractory Multiple Myeloma
Brief Title: Elotuzumab, Selinexor, and Dexamethasone for Relapsed Refractory Multiple Myeloma
Acronym: ESdRRMM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study collaborator -Karyopharm- is not doing Myeloma studies funding, so they let the study investigators know they are not funding the study anymore.
Sponsor: Tulane University School of Medicine (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-342
Record Dates: First submitted 2021-10-11; First posted 2021-12-28 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
Keywords: Multiple myeloma; Relapsed; Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — elotuzumab; selinexor; Dexamethasone

STUDY DESIGN:
Intervention Model Description: All patients enrolled in this clinical trial will receive the study drugs; elotuzumab, selinexor, and dexamethasone (ESd).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention arm (Experimental): This study employs a single, intervention arm or group, anticipated size of which is 18 patients, in which all enrolled subjects will receive the study drug, ESd.
  Interventions: Drug: Elotuzumab, Selinexor, and Dexamethasone (ESd)

INTERVENTIONS:
Drug: Elotuzumab, Selinexor, and Dexamethasone (ESd) — This is a single-arm, interventional, phase II clinical trial, in which the anticipated 18 enrolled patients will receive the trial drug, a combination of Elotuzumab, Selinexor, and Dexamethasone in monthly cycles. The study tests the theory of synergy between these drugs, as detailed in the study description above.

SUMMARY:
The food and drug administration (FDA) has approved the use of Selinexor, an oral, first-in class, exportin 1 (XPO1) inhibitor, in combination with low-dose dexamethasone in patients with triple-refractory (disease refractory to proteasome inhibitors (PI), immunomodulatory imid agents (IMiD), and anti-Cluster of Differentiation 38 (CD38) monoclonal antibodies (mAb)), or relapsed refractory multiple myeloma (RRMM). SLAMF7 (human Signaling Lymphocyte Activation Molecule Family 7) is a receptor that is present on immune cells, NK (Natural Killer) cells, and plasma cells. Elotuzumab, a mAb directed against the extracellular domain of SLAMF7, is used in combination with an IMiD and dexamethasone to treat RRMM. In this clinical trial, the investigators are proposing the addition of Elotuzumab to Selinexor and low-dose dexamethasone (ESd) in RRMM, previously treated with one or a combination of PI's, IMiD's, and anti-CD38 mAb.

DETAILED DESCRIPTION:
Selinexor reversibly inhibits nuclear export of tumor suppressor proteins (TSPs) resulting in a pro-apoptotic effect. In addition, previous studies found that selinexor alone or in combination with anti-PD-L1 (Programmed Death-Ligand 1) antibody significantly increased the frequency of natural killer cells on immunophenotypic analysis of splenocytes by flow cytometry. Elotuzumab activates NK cells through SLAMF7 and results in NK cell-mediated antibody dependent cellular toxicity (ADCC.) This clinical trial is designed on the premise that these two medications could have a synergistic effect resulting in a better clinical response in the treatment of RRMM.

The investigators will evaluate the ORR (overall response rate), CR (Complete Response), VGPR (Very Good Partial Response), PR (Partial Response) rates and the duration of response. Special consideration will be given to multiple myeloma patients with t(11;14) (q13;q32), given it is the most common chromosome translocation in multiple myeloma with early reported activity of Selinexor on BCR (Breakpoint Cluster Region Protein) inhibition. Finally, the investigators will evaluate the correlation between NK function and the response rate to possibly develop a predictive model of response rate to the combination based on NK activity measurements, pre, during, and post treatment. Quantitative testing includes the number of NK (CD3-, CD56/16+) cells, NK subsets (CD56bright to CD56dim ratio) and qualitative testing includes chromium release assay (using 51Cr) for cytotoxicity testing. In addition, the investigators will follow the response of African American patients to this regimen in an ancillary, ad hoc study given the under representation in the STORM (Selinexor Treatment of Refractory Myeloma) trial.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible to enroll in this study:

1. Age ≥ 18 years
2. Willing and able to provide written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of ≤ 2
4. Having measurable MM based on the modified International Myeloma Working Group (IMWG) guidelines, defined by at least one of the following: Serum M-protein

   ≥ 0.5 g/dL by serum electrophoresis (SPEP), urinary M-protein excretion ≥ 200 mg/24 hours by urine electrophoresis (UPEP), and free light chain (FLC) ≥ 100 mg/L, provided that the FLC ratio is abnormal.
5. Patients with non-secretory multiple myeloma will be included if they have 25% or more of plasmacytoma size progression or appearance of new plasmacytoma lesions.
6. Must have at least previously received ≥ 1 anti-MM regimens
7. More than 6 months have passed since an allogeneic transplant or 100 days since an autologous stem cell transplant, if patients had any
8. Adequate hepatic function within 28 days prior to C1D1:

   1. Total bilirubin < 1.5 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 × ULN), and
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (3) normal to<2 × ULN.
9. Calculated creatinine clearance (CrCl) >15 mL/min based on the Cockcroft and Gault formula.
10. Adequate hematopoietic function within 7 days prior to C1D1: total white blood cell (WBC) count ≥1500/mm3, absolute neutrophil count ≥1000/mm3, hemoglobin

    ≥8.5 g/dL and platelet count ≥75,000/mm3
    1. Patients receiving hematopoietic growth factor support, including erythropoietin, darbepoetin, granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), and platelet stimulators (eg, eltrombopag, romiplostim, or interleukin-11) must have at least a 2-week interval between growth factor support and the Screening assessments, but they may receive growth factor support during the study.
    2. Patients must have:

       * At least a 2-week interval from the last red blood cell (RBC) transfusion prior to the Screening hemoglobin assessment, and
       * At least a 1-week interval from the last platelet transfusion prior to the Screening platelet assessment.
11. Female patients of childbearing potential must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly
12. Effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not eligible to enroll in this study:

1. Has received selinexor or another XPO1 inhibitor previously.
2. Has any concurrent medical condition or disease (eg, uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.) that is likely to interfere with study procedures.
3. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to Cycle 1 Day 1 (C1D1). Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
4. Known intolerance, hypersensitivity, or contraindication to glucocorticoids.
5. Pregnant or breastfeeding females.
6. Life expectancy of <6 months
7. Major surgery within 6 weeks prior to C1D1.
8. Patients with active hepatitis B virus (HBV) are eligible if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 IU/mL.
9. Patients with untreated hepatitis C virus (HCV) are eligible if there is a documentation of negative viral load per institutional standard.
10. Patients with history of human immunodeficiency virus (HIV) are eligible if they have cluster of differentiation 4 (CD4+ )T-cell counts ≥350 cells/µL, negative viral load per institutional standard, and no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections in the last year.
11. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
12. Inability or unwillingness to take supportive medications such as anti-nausea and anti-anorexia agents as recommended by the National Cancer Comprehensive Network (NCCN) for antiemesis and anorexia/cachexia (palliative care).
13. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
14. Contraindication to any of the required concomitant drugs or supportive treatments.
15. Patients unwilling or unable to comply with the protocol including providing 24-hour urine samples for urine protein electrophoresis at the required time points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Response of relapsed refractory multiple myeloma (RRMM) patient to elotuzumab, selinexor, and dexamethasone (ESd). | 18-24 months.
  Calculate the Overall Response Rate (ORR) as the percentage of participants responding, as per the international working myeloma group (IMWG) criteria, mainly by following bone marrow plasma cell, serum, and urine monoclonal protein and free light chain production, by the date of study completion and on further, predetermined, follow up intervals of the study participants.

SECONDARY OUTCOMES:
Incidence of adverse events in RRMM patients treated with ESd. | 18-24 months.
  Will be assessed per the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 which is a standardized scale used to quantify the severity of chemotherapy-related adverse events, ranging from grade I, which is the mildest, to grade 4, which is the most severe, and grade 5, which is death.
Duration of Response (DOR) of RRMM patients to ESd. | 18-24 months.
  DOR is determined by the length of time in months from when measurement criteria for response were first met until the date of first recurrence, progressive disease [PD] or death. The unit of measure is month.
Overall Survival (OS) of RRMM patients treated with ESd. | 18-24 months.
  The investigators will determine the OS to ESd in patients with MM refractory to at least one prior line of treatment. The unit of measure is month.

CONTACTS AND LOCATIONS:
Overall Officials: Hana Safah, MD, Principal Investigator — Tulane University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reversal of immune tolerance and increased anti tumoral immune response in a mouse model of CNS B cell lymphoma after combined XPO1 and BCR inhibition Marta Crespo, Isabel Jiménez, Júlia Carabia, Sabela Bobillo, Pau Abrisqueta, Carles Palacio, Juan Camilo Nieto, Joan Boix, Cecilia del Carmen Carpio, Josep Castellví, Joan Seoane and Francesc Bosch Cancer Res July 1 2018 (78) (13 Supplement) 4568; DOI: 10.1158/1538-7445.AM2018-4568
- [Result] Farren MR, Hennessey RC, Shakya R, Elnaggar O, Young G, Kendra K, Landesman Y, Elloul S, Crochiere M, Klebanov B, Kashyap T, Burd CE, Lesinski GB. The Exportin-1 Inhibitor Selinexor Exerts Superior Antitumor Activity when Combined with T-Cell Checkpoint Inhibitors. Mol Cancer Ther. 2017 Mar;16(3):417-427. doi: 10.1158/1535-7163.MCT-16-0498. Epub 2017 Feb 1. PMID 28148715
- [Result] An G, Xu Y, Shi L, Zou D, Deng S, Sui W, Xie Z, Hao M, Chang H, Qiu L. t(11;14) multiple myeloma: a subtype associated with distinct immunological features, immunophenotypic characteristics but divergent outcome. Leuk Res. 2013 Oct;37(10):1251-7. doi: 10.1016/j.leukres.2013.06.020. Epub 2013 Aug 5. PMID 23927993
- [Result] Chari A, Vogl DT, Gavriatopoulou M, Nooka AK, Yee AJ, Huff CA, Moreau P, Dingli D, Cole C, Lonial S, Dimopoulos M, Stewart AK, Richter J, Vij R, Tuchman S, Raab MS, Weisel KC, Delforge M, Cornell RF, Kaminetzky D, Hoffman JE, Costa LJ, Parker TL, Levy M, Schreder M, Meuleman N, Frenzel L, Mohty M, Choquet S, Schiller G, Comenzo RL, Engelhardt M, Illmer T, Vlummens P, Doyen C, Facon T, Karlin L, Perrot A, Podar K, Kauffman MG, Shacham S, Li L, Tang S, Picklesimer C, Saint-Martin JR, Crochiere M, Chang H, Parekh S, Landesman Y, Shah J, Richardson PG, Jagannath S. Oral Selinexor-Dexamethasone for Triple-Class Refractory Multiple Myeloma. N Engl J Med. 2019 Aug 22;381(8):727-738. doi: 10.1056/NEJMoa1903455. PMID 31433920